CLINICAL TRIAL: NCT04774094
Title: A SINGLE ARM, OPEN-LABEL, MULTI-CENTER, INTERVENTIONAL STUDY EVALUATING THE EFFICACY AND SAFETY OF CEFTAZIDIME-AVIBACTAM (CAZ-AVI) IN CHINESE ADULTS WITH HAP (INCLUDING VAP)
Brief Title: Efficacy and Safety of Ceftazidime-Avibactam (CAZ-AVI) in Chinese Participants With HAP (Including VAP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C3591026
Record Dates: First submitted 2021-02-05; First posted 2021-03-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Hospital-Acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAZ-AVI (Experimental)
  Interventions: Drug: Zavicefta, Ceftazidime-Avibactam

INTERVENTIONS:
Drug: Zavicefta, Ceftazidime-Avibactam — Participants will receive CAZ-AVI (2000 mg of ceftazidime and 500 mg of avibactam) administered by IV infusion in a volume of 100 mL at a constant rate over 2 hours.

SUMMARY:
This is a prospective, single arm, open-label, multi-center clinical study evaluating the effectiveness and safety of CAZ-AVI in participants with HAP (including VAP), who have initiated treatment with CAZ-AVI in an inpatient hospital setting. The duration of antibiotic treatment with the CAZ-AVI is 7-14 days. Participants must receive intravenously (IV) CAZ-AVI in the hospital for at least 7 full days. There are no formal hypothesis tests planned for this study. The number and percent of participants having clinical cure, failure, and indeterminate at TOC visit in the cMITT analysis population will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 and ≤90 years of age.
* Onset of symptoms ≥48 hours after admission or <7 days after discharge from an inpatient acute or chronic care facility.
* New or worsening infiltrate on chest X-ray obtained within 48 hours prior to screening.
* Participants have systemic signs and respiratory signs or symptoms of HAP/VAP

Exclusion Criteria:

* Other medical or psychiatric condition may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Participant is expected to require a treatment course for HAP longer than 14 days.
* The total duration of antibiotic exposure for antibiotics whose administration begins in the 48 hours is longer than 24 hours.
* Previous administration with an investigational drug within 30 days or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* Acute Physiology and Chronic Health Evaluation (APACHE) II score >30 or <10 using the most recent available data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- China (54):
  - Fuyang People's Hospital, Fuyang, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Zhongshan Hospital Xiamen University, Xiamen, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - ZhuJiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Second People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - The Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Sanya People's Hospital, Sanya, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Luoyang Central Hospital, Luoyang, Henan
  - NanYang central hospital, Nanyang, Henan
  - NanYang First people's hospital, Nanyang, Henan
  - Henan provincial people's hospital, Zhengzhou, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Yueyang People's Hospital, Yueyang, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - The First People's Hospital of Lianyungang City, Lianyungang, Jiangsu
  - Taizhou People's Hospital, Taizhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Chengdu Xinhua Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - The First Hospital of Kunming, Kunming, Yunnan
  - Dongyang People's Hospital, Dongyang, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The 2nd Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - Seventh Medical Center, The General Hospital of People's Liberation Army, Beijing
  - Shanghai Fifth People's Hospital, Fudan University, Shanghai
  - Zhongshan Hospital Xiamen University, Xiamen

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3591026

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 235 Chinese adult participants with hospital acquired pneumonia (HAP) [including ventilator-associated pneumonia {VA}] were enrolled.
Groups:
- Ceftazidime-Avibactam (CAZ-AVI): Participants received CAZ-AVI (Zavicefta), 2.5 grams (g) [ceftazidime 2g + avibactam 0.5g], intravenously (IV) as 2 hours infusion every 8 hours for a minimum of 7 days and a maximum of 14 days. Participants were followed up to maximum of 32 days after the last dose of study intervention.
Period: Overall Study
Arm/Group | Ceftazidime-Avibactam (CAZ-AVI)
Started | 235
Completed | 191
Not Completed | 44
Not completed — Other | 2
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 7
Not completed — Lack of Efficacy | 5
Not completed — Death | 17
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS) included all participants who had taken at least 1 dose of study intervention.
Groups:
- CAZ-AVI 1: Participants received CAZ-AVI (Zavicefta), 2.5 g (ceftazidime 2g + avibactam 0.5g), IV as 2 hours infusion every 8 hours for a minimum of 7 days and a maximum of 14 days. Participants were followed up to maximum of 32 days after the last dose of study intervention.
Arm/Group | CAZ-AVI 1
Number analyzed (Participants) | 235
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 235
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 235
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Cure at Test of Cure (TOC) Visit: Clinical Modified Intent-to-Treat (cMITT) Population
Description: Clinical cure: participants were considered to be a success for clinical response at TOC visit if the participants were not a clinical failure at end of treatment (EOT), and the participants were alive and all signs and symptoms of pneumonia were resolved or improved to an extent that no antibacterial therapy for HAP was taken between EOT and TOC inclusive. Gram negative is abbreviated as gram -ve and gram positive as gram +ve.
Time Frame: TOC visit: any day from Day 21 to 25
Population: cMITT: MITT subset and participants whose baseline respiratory or blood culture showed gram -ve pathogens with or without concomitant gram +ve pathogens (excluding those with gram -ve pathogens unexpected to respond to either study drug [participants with only monomicrobial gram -ve infection: any Acinetobacter species/ Legionella species/ Stenotrophomonas maltophilia/ Elizabethkingia meningoseptica]) or in whom no etiologic pathogens identified from respiratory or blood culture at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- CAZ-AVI: Participants with HAP received CAZ-AVI, 2.5 g, IV as 2 hours infusion every 8 hours for a maximum of 14 days.
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 209
Percentage of participants | 62.7 [56.0 to 69.0]

2. Secondary Outcome: Percentage of Participants With Clinical Cure at EOT Visit: cMITT Population
Description: Clinical cure: participants were considered to be a success for clinical response at EOT visit if the participants were alive and all signs and symptoms of pneumonia were resolved or improved such that all antibacterial therapies for HAP/ VAP were stopped. No antibacterial therapy other than those outlined by the protocol was administered for HAP prior to EOT.
Time Frame: EOT visit: within 24 hours after the completion of the last infusion of study intervention (study treatment was a minimum of 7 days and maximum of 14 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 209
Percentage of participants | 75.1 [68.9 to 80.6]

3. Secondary Outcome: Percentage of Participants With Clinical Cure at EOT and TOC Visit: Microbiological Modified Intent-to-Treat (mMITT) Population
Description: Clinical cure at EOT: participants were considered to be a success for clinical response at EOT visit if the participants were alive and all signs and symptoms of pneumonia were resolved or improved such that all antibacterial therapies for HAP/VAP were stopped. No antibacterial therapy other than those outlined by the protocol was administered for HAP prior to EOT. Clinical cure at TOC: participants were considered to be a success for clinical response at TOC visit if the participants were not a clinical failure at EOT, and the participants were alive and all signs and symptoms of pneumonia were resolved or improved to an extent that no antibacterial therapy for HAP was taken between EOT and TOC inclusive.
Time Frame: EOT visit: within 24 hours after the completion of the last infusion of study intervention (study treatment was a minimum of 7 days and maximum of 14 days); TOC visit: any day from Day 21 to 25
Population: mMITT:MITT subset and participants with proper respiratory culture (RC) showing gram-ve pathogens,excluding participants unexpected to respond to CAZ-AVI (participants with only monomicrobial gram-ve infections:any Acinetobacter species/Legionella species/Stenotrophomonas maltophilia/Elizabethkingia meningoseptica).If baseline RC unavailable or didn't identify respiratory pathogen, but gram-ve organism causing pneumonia was identified from baseline blood cultures,participant qualified for mMITT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 80
Percentage of participants
  EOT visit | 70.0 [59.4 to 79.2]
  TOC visit | 57.5 [46.6 to 67.9]

4. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiological Response at the EOT and TOC Visits: mMITT Population
Description: For participants from whom only 1 causative pathogen is isolated, the overall microbiological response assessment was based on the microbiological response assessment for that pathogen. For participants from whom more than 1 baseline pathogen was isolated, the overall microbiological response assessment was "favorable" only if the microbiological response assessment for each of the baseline pathogens isolated was "favorable". Favorable microbiological response included eradication (an adequate source specimen demonstrated absence of the original baseline pathogen) and presumed eradication (an adequate source specimen was not available to culture and the participant was assessed as a clinical cure). In this outcome measure percentage of participants with favorable per-participant microbiological response are recorded.
Time Frame: as for outcome 3
Population: mMITT:MITT subset and participants with proper RC showing gram-ve pathogens,excluding participants unexpected to respond to CAZ-AVI (participants with only monomicrobial gram-ve infections:any Acinetobacter species/Legionella species/Stenotrophomonas maltophilia/Elizabethkingia meningoseptica).If baseline RC unavailable or didn't identify respiratory pathogen, but gram-ve organism causing pneumonia was identified from baseline blood cultures,participant qualified for mMITT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 80
Percentage of participants
  EOT visit | 77.5 [67.5 to 85.6]
  TOC visit | 51.3 [40.4 to 62.0]

5. Secondary Outcome: Percentage of Participants With Favorable Per-Pathogen Microbiological Response at the EOT and TOC Visits: mMITT Population
Description: Favorable microbiological response included eradication (an adequate source specimen demonstrated absence of the original baseline pathogen) and presumed eradication (an adequate source specimen was not available to culture and the participant was assessed as a clinical cure). In this outcome measure percentage of participants with favorable per-pathogen microbiological response are recorded.
Time Frame: as for outcome 3
Population: mMITT analysis set evaluated. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies number of participants in mMITT analysis set evaluable for specified pathogens and visits.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 80
Percentage of participants
  EOT visit: Enterobacter cloacae: number analyzed (Participants) | 3
  EOT visit: Enterobacter cloacae | 33.3 [3.9 to 82.3]
  EOT visit: Escherichia coli: number analyzed (Participants) | 5
  EOT visit: Escherichia coli | 100 [62.1 to 100]
  EOT visit: Klebsiella aerogenes: number analyzed (Participants) | 5
  EOT visit: Klebsiella aerogenes | 80.0 [37.1 to 97.7]
  EOT visit: Klebsiella pneumoniae: number analyzed (Participants) | 49
  EOT visit: Klebsiella pneumoniae | 77.6 [64.5 to 87.4]
  EOT visit: Klebsiella variicola: number analyzed (Participants) | 1
  EOT visit: Klebsiella variicola | 100 [14.7 to 100]
  EOT visit: Morganella morganii: number analyzed (Participants) | 1
  EOT visit: Morganella morganii | 100 [14.7 to 100]
  EOT visit: Proteus mirabilis: number analyzed (Participants) | 3
  EOT visit: Proteus mirabilis | 100 [46.4 to 100]
  EOT visit: Proteus vulgaris: number analyzed (Participants) | 1
  EOT visit: Proteus vulgaris | 100 [14.7 to 100]
  EOT visit: Providencia rettgeri: number analyzed (Participants) | 1
  EOT visit: Providencia rettgeri | 100 [14.7 to 100]
  EOT visit: Providencia stuartii: number analyzed (Participants) | 1
  EOT visit: Providencia stuartii | 100 [14.7 to 100]
  EOT visit: Serratia marcescens: number analyzed (Participants) | 1
  EOT visit: Serratia marcescens | 100 [14.7 to 100]
  EOT visit: Acinetobacter baumannii: number analyzed (Participants) | 7
  EOT visit: Acinetobacter baumannii | 71.4 [35.2 to 93.5]
  EOT visit: Haemophilus influenzae: number analyzed (Participants) | 4
  EOT visit: Haemophilus influenzae | 100 [55.5 to 100]
  EOT visit: Moraxella catarrhalis: number analyzed (Participants) | 1
  EOT visit: Moraxella catarrhalis | 0 [0.0 to 85.3]
  EOT visit: Pseudomonas aeruginosa: number analyzed (Participants) | 16
  EOT visit: Pseudomonas aeruginosa | 75.0 [50.9 to 90.9]
  EOT visit: Stenotrophomonas maltophilia: number analyzed (Participants) | 2
  EOT visit: Stenotrophomonas maltophilia | 50.0 [6.1 to 93.9]
  EOT visit: Enterococcus faecium: number analyzed (Participants) | 1
  EOT visit: Enterococcus faecium | 100 [14.7 to 100]
  EOT visit: Staphylococcus aureus: number analyzed (Participants) | 7
  EOT visit: Staphylococcus aureus | 57.1 [23.5 to 86.1]
  EOT visit: Staphylococcus hominis: number analyzed (Participants) | 1
  EOT visit: Staphylococcus hominis | 100 [14.7 to 100]
  TOC visit: Enterobacter cloacae: number analyzed (Participants) | 3
  TOC visit: Enterobacter cloacae | 33.3 [3.9 to 82.3]
  TOC visit: Escherichia coli: number analyzed (Participants) | 5
  TOC visit: Escherichia coli | 100 [62.1 to 100]
  TOC visit: Klebsiella aerogenes: number analyzed (Participants) | 5
  TOC visit: Klebsiella aerogenes | 80.0 [37.1 to 97.7]
  TOC visit: Klebsiella pneumoniae: number analyzed (Participants) | 49
  TOC visit: Klebsiella pneumoniae | 53.1 [39.2 to 66.5]
  TOC visit: Klebsiella variicola: number analyzed (Participants) | 1
  TOC visit: Klebsiella variicola | 100 [14.7 to 100]
  TOC visit: Morganella morganii: number analyzed (Participants) | 1
  TOC visit: Morganella morganii | 100 [14.7 to 100]
  TOC visit: Proteus mirabilis: number analyzed (Participants) | 3
  TOC visit: Proteus mirabilis | 66.7 [17.7 to 96.1]
  TOC visit: Proteus vulgaris: number analyzed (Participants) | 1
  TOC visit: Proteus vulgaris | 100 [14.7 to 100]
  TOC visit: Providencia rettgeri: number analyzed (Participants) | 1
  TOC visit: Providencia rettgeri | 100 [14.7 to 100]
  TOC visit: Providencia stuartii: number analyzed (Participants) | 1
  TOC visit: Providencia stuartii | 100 [14.7 to 100]
  TOC visit: Serratia marcescens: number analyzed (Participants) | 1
  TOC visit: Serratia marcescens | 100 [14.7 to 100]
  TOC visit: Acinetobacter baumannii: number analyzed (Participants) | 7
  TOC visit: Acinetobacter baumannii | 42.9 [13.9 to 76.5]
  TOC visit: Haemophilus influenzae: number analyzed (Participants) | 4
  TOC visit: Haemophilus influenzae | 100 [55.5 to 100]
  TOC visit: Moraxella catarrhalis: number analyzed (Participants) | 1
  TOC visit: Moraxella catarrhalis | 0 [0.0 to 85.3]
  TOC visit: Pseudomonas aeruginosa: number analyzed (Participants) | 16
  TOC visit: Pseudomonas aeruginosa | 37.5 [17.4 to 61.7]
  TOC visit: Stenotrophomonas maltophilia: number analyzed (Participants) | 2
  TOC visit: Stenotrophomonas maltophilia | 0 [0.0 to 66.7]
  TOC visit: Enterococcus faecium: number analyzed (Participants) | 1
  TOC visit: Enterococcus faecium | 100 [14.7 to 100]
  TOC visit: Staphylococcus aureus: number analyzed (Participants) | 7
  TOC visit: Staphylococcus aureus | 42.9 [13.9 to 76.5]
  TOC visit: Staphylococcus hominis: number analyzed (Participants) | 1
  TOC visit: Staphylococcus hominis | 100 [14.7 to 100]

6. Secondary Outcome: Percentage of Participants With Clinical Cure at the EOT and TOC Visits in Participants With Gram-negative Baseline Pathogens Resistant to Ceftazidime: mMITT Population
Description: as for outcome 3
Time Frame: as for outcome 3
Population: mMITT analysis set evaluated. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure, i.e. participants in mMITT analysis set that with gram-negative baseline pathogens resistant to ceftazidime.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 30
Percentage of participants
  EOT visit | 63.3 [45.5 to 78.7]
  TOC visit | 53.3 [35.9 to 70.2]

7. Secondary Outcome: Percentage of Participants With Favorable Per-Participant Microbiologic Response at the EOT and TOC Visits in Participants With Gram-negative Baseline Pathogens Resistant to Ceftazidime: mMITT Population
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 30
Percentage of participants
  EOT visit | 73.3 [55.9 to 86.5]
  TOC visit | 46.7 [29.8 to 64.1]

8. Secondary Outcome: Percentage of Participants With Death Due to Any Cause at the TOC Visit and at Day 28 Visit: cMITT Population
Time Frame: TOC visit: any day from Day 21 to 25; Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 209
Percentage of participants
  TOC visit | 5.7 [3.2 to 9.5]
  Day 28 visit | 5.7 [3.2 to 9.5]

9. Secondary Outcome: Percentage of Participants With Death Due to Any Cause at the TOC Visit and at Day 28 Visit: mMITT Population
Time Frame: TOC visit: any day from Day 21 to 25; Day 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 80
Percentage of participants
  TOC visit | 7.5 [3.2 to 14.8]
  Day 28 visit | 7.5 [3.2 to 14.8]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and all non-SAEs that occurred in the study. TEAEs were AEs between first dose of study treatment and up to 32 days post last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to 32 days after last dose of CAZ-AVI (maximum up to 46 days; maximum treatment duration was of 14 days)
Population: SAS included all participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 235
Participants | 204

11. Secondary Outcome: Number of Participants With Clinically Significant Post-Baseline Laboratory Test Abnormalities
Description: Hematology: Hemoglobin (Hg), hematocrit, erythrocytes: less than (<)0.8*lower limit of normal (LLN) & change (chg) more than (>)20% decrease (dec); platelets: <0.65*LLN & chg >50% dec &, >1.5* upper limit of normal (ULN) & chg >100% increase (inc); leukocytes: <0.65*LLN & chg >60% dec &, >1.6*ULN & chg >100% inc; lymphocytes, <0.25*LLN & chg >75% dec; neutrophils: <0.65*LLN & chg >75% dec &, >1.6*ULN & chg >100% inc; basophils, monocytes: >4.0* ULN & chg >300% inc. Clinical chemistry: bilirubin: >2.0*ULN & chg >150% inc; aspartate aminotransferase (AT) & Alanine AT: >3.0*ULN & chg >200% inc; alkaline phosphatase <0.5*LLN & chg >80% dec & >2.0*ULN & chg >100% inc; creatinine: >2.0*ULN & >chg 100% inc; sodium: <0.85*LLN & chg >10% dec & >1.1*ULN & chg >10% inc; potassium & chloride: <0.8*LLN & chg >20% dec & >1.2*ULN & chg >20% dec; calcium: <0.7*LLN & chg >30% dec & bicarbonate: <0.7*LLN & chg >40% dec. Clinical significance was judged by investigator.
Time Frame: Day 1 up to 32 days after last dose of CAZ-AVI (maximum up to 46 days; maximum treatment duration was of 14 days)
Population: SAS included all participants who had taken at least 1 dose of study intervention. Here "Number of Participants Analyzed" includes number of participants evaluable for laboratory abnormalities.
Measure: Count of Participants; unit: Participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 234
Participants | 102

12. Secondary Outcome: Number of Participants With Vital Signs Data According to Pre-defined Criteria
Description: Vital signs included diastolic blood pressure (millimeters of mercury [mmHg]); pulse rate (beats per minute [bpm]) and systolic blood pressure (mmHg). Pre-defined criteria: Diastolic blood pressure: Value <50 mmHg, Diastolic blood pressure: Change more than or equal to (>=) 20 mmHg increase, Diastolic blood pressure: Change >= 20 mmHg decrease, Pulse rate: Value <40 bpm, Pulse rate: Value >120 bpm, Systolic blood pressure: Value <90 mmHg, Systolic blood pressure: Change >= 30 mmHg increase, Systolic blood pressure: Change >= 30 mmHg decrease. One participant could have more than one vital sign abnormality.
Time Frame: Day 1 up to 32 days after last dose of CAZ-AVI (maximum up to 46 days; maximum treatment duration was of 14 days)
Population: SAS included all participants who had taken at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | CAZ-AVI
Number analyzed (Participants) | 235
Participants
  Diastolic blood pressure: <50 mmHg | 18
  Diastolic blood pressure: Change >=20 mmHg increase | 72
  Diastolic blood pressure: Change >= 20 mmHg decrease | 54
  Pulse rate: Value <40 bpm | 1
  Pulse rate: Value >120 bpm | 31
  Systolic blood pressure: Value <90 mmHg | 11
  Systolic blood pressure: Change >= 30 mmHg increase | 61
  Systolic blood pressure: Change >= 30 mmHg decrease | 64

ADVERSE EVENTS:
Time Frame: Day 1 up to 32 days after last dose of CAZ-AVI (maximum up to 46 days; maximum treatment duration was of 14 days)
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Non-SAES are reported at 5% threshold.
Groups:
- CAZ-AVI: Participants received CAZ-AVI (Zavicefta), 2.5 g (ceftazidime 2g + avibactam 0.5g), IV as 2 hours infusion every 8 hours for a minimum of 7 days and a maximum of 14 days. Participants were followed up to maximum of 32 days after the last dose of study intervention.
Arm/Group | CAZ-AVI
All-Cause Mortality (participants affected / at risk) | 17/235
Serious Adverse Events (participants affected / at risk) | 35/235
Other Adverse Events (participants affected / at risk) | 43/235
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAZ-AVI (N=235)
Cardiac arrest (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Effusion (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Liver injury (Hepatobiliary disorders) | 2
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1
Fungaemia (Infections and infestations) | 1
Intracranial infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia aspiration (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Puncture site infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Brain herniation (Injury, poisoning and procedural complications) | 2
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2
Subdural effusion (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CAZ-AVI (N=235)
Diarrhoea (Gastrointestinal disorders) | 17
Hepatic function abnormal (Hepatobiliary disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT04774094/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/94/NCT04774094/SAP_001.pdf